CLINICAL TRIAL: NCT00993395
Title: A Comprehensive Peer Mentor-based Disease Management Program for Medically Complex Substance Users
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Healthways, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00020931
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Substance Addiction
Keywords: addiction; peer mentor; adherence
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peer Mentor Intervention (Experimental): peer mentor-based disease management focusing on three domains: medical care, recovery, and social stabilization
  Interventions: Behavioral: peer mentor-based disease management

INTERVENTIONS:
Behavioral: peer mentor-based disease management — peer mentor-based disease management focused on three domains: medical care, recovery, and social stabilization

SUMMARY:
Substance-using adults are admitted to hospital for medical complication from their drug and alcohol use at very high rates; yet, their care is often defined by low rates of referral to addiction treatment programs and recidivism. In 1997, we instituted an integrated medical-substance use treatment program at Johns Hopkins, the First Step Day Hospital, designed for intensive post-acute care of previously hospitalized substance using adults. We have shown that patients with dual diagnoses admitted to First Step more often complete their course of medical care and stay in recovery longer than patients not admitted to First Step.(1;2) On discharge from First Step, patients are medically stable and drug-free. Their substance abuse care is transferred to an out-patient substance abuse treatment facility and their medical care is transferred to their primary care provider. Unfortunately, many patients are lost to follow-up during this transition. We believe that a peer mentor-based disease management program (PM) can provide continuity of care that begins in First Step and continues after discharge thereby increasing the proportion of patients who remain in treatment for their addiction and medical conditions. Peer mentors are persons from the target community who have been in recovery for 5 or more years. In cooperation with patients and providers, peer mentors improve the integration of care, quality of care, and access to healthcare services. This pilot study will test the effectiveness of a peer mentor-based disease management program. The specific aims are to compare the impact of the PM intervention verses enhanced usual care on outcomes in three domains (1) medical/psychiatric health status, (2) addiction recovery, and (3) social resource acquisition. If successful, this study will provide evidence supporting a larger randomized controlled trial of the impact of field workers on post-acute care among patients with dual diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to an intensive day hospital focused on medically complex substanse users are eligible for enrolment

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
adherence to first prescription refill after discharge | 60 days

SECONDARY OUTCOMES:
Adherence to first medical appointment | 60 days
Rate of readmission and emergency department visits | 3 years
Length of stay in a recovery program | 1 year
Number of days without substance use | 3 years
Acquisition of medical insurance | 1 year
acquisition of long-term housing | 3 years
Acquisition of financial support | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States